CLINICAL TRIAL: NCT04432272
Title: ANTIBODY-LEVEL BASED ANALYSIS OF COVID-19 CONVALESCENT SERUM (ABACCuS)
Acronym: ABACCuS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The EUA for CCP was updated by FDA, stipulating that only high titer units be used. This study required untitered units. The study became infeasible
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Matthew Sims, MD, PhD, Director Infectious Disease Research, Beaumont Health; Professor of Internal Medicine and Foundational Medical Studies, OUWB School of Medicine, Corewell Health East
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-198
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Severe Acute Respiratory Syndrome (SARS); Coronavirus Infections
Keywords: therapeutic treatment; COVID-19 convalescent plasma; anti-SARS-CoV-2 antibody; IgA; IgG; COVID-19 pandemic
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: Prospective, single health system, non-randomized, open-label study.
Masking Description: No parties blinded as to receipt of study article. Participant, care provider and investigator blinded to actual antibody concentration in unit of plasma provided.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Hospitalized COVID-19 patients ages ≥18 years with respiratory symptoms, requiring >6 L of oxygen to maintain oxygen saturation >92%. Patient may not require intubation, and may be admitted for no longer than 14 days.
  Interventions: Biological: COVID-19 convalescent plasma
- Group B (Experimental): Hospitalized COVID-19 patients ages ≥18 years requiring intubation.
  Interventions: Biological: COVID-19 convalescent plasma

INTERVENTIONS:
Biological: COVID-19 convalescent plasma — Participants will receive 1 unit of convalescent plasma procured from donors who have: 1) been symptom free for 14 days and screen negative via nasopharyngeal swab or 2) symptom free for at least 28 days or 3) individuals who have never had symptoms of COVID-19 but were found to have elevated anti-SARS-CoV-2 IgG by a serology test deemed to be of acceptable quality and fitting the current guidance by the FDA. Participants, clinicians, investigators and outcomes assessors will be blinded to the amount of anti-SARS-CoV-2 IgA and IgG present in each unit

SUMMARY:
The goal of this study is to evaluate the safety and effectiveness of Coronavirus-90 (COVID-19) convalescent plasma for the treatment of COVID-19. Plasma is the liquid part of blood that is left when all the blood cells have been removed. Convalescent means it is taken from people who were infected with COVID-19 and recovered. The use of this blood product to treat COVID-19 is investigational, which means the U.S. Food and Drug Administration has not yet approved it to be sold commercially. This is a human blood product collected by licensed blood banks. Donors of COVID-19 convalescent plasma must meet all standard blood donor criteria and must also meet all criteria set by the FDA for being a donor of COVID-19 convalescent plasma.

A total of 500 patients will take part in the study at 8 hospitals within Beaumont. Similar studies are being done at other centers, but they are not directly related to this study.

Participants will be assigned to a study group depending on how sick they are.

* Group A: Those who require more than 6 liters (L) of supplemental oxygen but are not on a ventilator
* Group B: Those who require a ventilator to preserve their life.

Both groups will receive one unit (approximately 200ml or just under 1 cup) of COVID convalescent plasma. The transfusion will be given over about 30 minutes via an IV. Blood samples will be taken prior to and one hour after the transfusion to measure participant antibodies against Severe Acute Respiratory Syndrome-Coronavirus 2 (SARS-CoV-2) and a nasopharyngeal swab (deep in the nostril) will be taken to test for presence of the SARS-CoV-2 virus. One hour after the transfusion a blood sample will be taken to measure antibody levels to determine if the plasma caused the antibody level to rise. Similarly, blood samples will be taken to measure antibodies against SARS-CoV-2 and a nasopharyngeal swab will be taken to test for presence of the SARS-CoV-2 virus 1, 3 and every 7 days after the transfusion while the participant is in the hospital The participant's final health status will be determined on day 28. Hospital records will be monitored for 90 days after discharge to determine if the participant is readmitted to the hospital.

DETAILED DESCRIPTION:
This trial will evaluate the efficacy and safety of SARS-CoV-2 convalescent plasma as treatment for confirmed COVID-19 respiratory disease (as defined in the inclusion criteria). Participants in both group A and group B will receive COVID-19 convalescent plasma. Group A will include hospitalized COVID-19 patients ages ≥18 years with respiratory symptoms, requiring >6 L of oxygen to maintain O2 saturation >92%. Patient may not require intubation, and may be admitted for no longer than 14 days. Group B will include hospitalized COVID-19 patients ages ≥18 years requiring intubation. Patients may be enrolled in group A within 14 days of admission to the hospital and may be enrolled in group B at any time after intubation. A total of 300 eligible subjects with significant oxygen requirements and 200 eligible subjects who require intubation will be included in the study. They will receive convalescent plasma from either a patient who has recovered from COVID-19 or from an asymptomatic carrier with confirmed Immunoglobulin-G (IgG) antibodies against SARS-CoV-2. Subjects will not be randomized. The amount of anti-SARS-CoV-2 IgG and Immunoglobulin-A (IgA) antibodies in any unit of plasma will not be known when the unit is assigned to the patient. This will allow us to examine the relationship between the amount of anti-SARS-CoV-2 antibody and outcomes. Analysis will be based on measurement of optical density of the IgG level in the unit of plasma the patient is randomly supplied by the blood bank. While investigators and patients will be aware the patient is receiving a unit of COVID-19 convalescent plasma, both the investigators and the patients will be blinded to the antibody content of that unit.

COVID-19 convalescent plasma (1 unit; ~200mL) will be produced by a blood bank licensed to produce plasma using standard screening and safety procedures. The product may be procured from patients who have: 1) been symptom free for 14 days and screen negative via nasopharyngeal swab or 2) symptom free for at least 28 days or 3) individuals who have never had symptoms of COVID-19 but were found to have elevated anti-SARS-CoV-2 IgG by a serology test deemed to be of acceptable quality and fitting the current guidance by the FDA.

Participants at the eight Michigan hospitals comprising the Beaumont Health system may be eligible to participate. Study oversight and coordination will occur centrally, from the Infectious Disease Research Department at Beaumont's Royal Oak campus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older.
* Hospitalized with confirmed COVID-19 infection via COVID-19 SARS-CoV-2 Reverse-transcription polymerase chain reaction (RT-PCR) testing.
* Symptoms consistent with COVID-19 infection (fever, acute onset cough, shortness of breath) at time of screening.
* Patient requires >6 L nasal cannula oxygen (Group A) or intubated (Group B).
* Patient (or their legal authorized representative) is willing and able to provide written informed consent and comply with all protocol requirements.

Exclusion Criteria:

* For patients in Group A admitted for >14 days
* Female subjects with positive pregnancy test, breastfeeding, or planning to become --pregnant or breastfeed during the study period.
* Receipt of pooled immunoglobulin in past 30 days.
* Contraindication to transfusion or history of prior reactions to transfusion blood products.
* Patients currently undergoing cancer treatment or those who are presently immunocompromised.
* Patient who in the opinion of the investigator will not be a good study candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sims, MD PhD, Principal Investigator — Beaumont Health
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 43 | 28
Completed | 43 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 43 | 28 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.95 (10.37) | 62.83 (13.53) | 68.96 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 30 | 19 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 40 | 26 | 66
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 41 | 20 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 43 | 28 | 71

OUTCOME MEASURES:

1. Primary Outcome: Avoidance of Intubation at 28 Days (Group A)
Description: Count of group A participants (non-intubated participants requiring >6 L supplemental oxygen to maintain oxygen saturation >92% at time of study entry and who are admitted <14 days) who remain un-intubated
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A
Number analyzed (Participants) | 43
Participants | 26

2. Primary Outcome: Mortality (Group B)
Description: Count of group B participants (participants who are intubated at study entry) who die
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group B
Number analyzed (Participants) | 28
Participants | 17

3. Secondary Outcome: Cardio-circulatory Arrest
Description: Count of participants who experienced cardio-circulatory arrest
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 28
Participants | 13 | 13

4. Secondary Outcome: Patient Outcome at 28 Days
Description: Patient Outcome as assessed on a 7-point ordinal scale, where 1= Not hospitalized, no limitations on activities, 2 =Not hospitalized, limitation on activities, 3= Hospitalized, not requiring supplemental oxygen, 4 =Hospitalized, requiring supplemental oxygen , 5 = Hospitalized, on non-invasive ventilation or high flow oxygen devices, 6 = Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO), 7=Deceased. A lower number indicates a better outcome
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 28
Participants
  1= Not hospitalized, no limitations on activities | 3 | 0
  2 =Not hospitalized, limitation on activities | 12 | 4
  3= Hospitalized, not requiring supplemental oxygen | 0 | 0
  4 =Hospitalized, requiring supplemental oxygen | 3 | 1
  5 = Hospitalized, on non-invasive ventilation or high flow oxygen devices | 2 | 1
  6 = Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | 2 | 5
  7=Deceased | 21 | 17

5. Secondary Outcome: Renal Failure
Description: Count of participants who develop or experience worsened renal failure as defined by RIFLE criteria, a 5-point scale where the categories are labeled: Risk-Injury-Failure-Loss-End stage renal disease, with Risk being the least severe and End stage renal disease being the most severe. The criteria for determination of stage are factors of serum creatinine and urine output. Numbers of participants worsening one or more RIFLE stages will be reported.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 28
Participants | 2 | 7

6. Secondary Outcome: Liver Failure
Description: Count of participants who develop or experience worsened liver failure as measured by elevation of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels to 5x the upper limit of normal or significant worsening of current liver failure with rise in transaminases of >25%
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 28
Participants | 1 | 1

7. Secondary Outcome: Cytokine Storm
Description: Count of participants who develop cytokine storm as measured by elevated markers of inflammation (elevated D-dimer, hypofibrinogenemia, hyperferritinemia), evidence of acute respiratory distress syndrome (ARDS) measured by imaging findings and mechanical ventilator requirements, and/or continuous fever (≥ 38.1 ° Celsius unremitting)
Time Frame: 28 days
Population: Data not available for 10 Group A participants and 8 group B participants
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 33 | 20
Participants | 9 | 5

8. Secondary Outcome: Respiratory Support
Description: Count of participants who require respiratory support in each of the following categories: nasal cannula, high flow nasal canula, non-rebreather mask, continuous positive airway pressure (CPAP), bilevel positive airway pressure (BIPAP), or intubation. Patients may receive more than one type of support during their hospital stay.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 28
Participants
  Ventilator | 19 | 27
  Coldflow | 1 | 0
  CPAP | 11 | 2
  BiPAP | 25 | 4
  Non-rebreather mask | 19 | 3
  Nasal cannula | 27 | 8
  High flow nasal cannula | 37 | 7

9. Secondary Outcome: Vasopressor Medication Support
Description: Count of participants who received pressor drugs, as ordered by treating physicians
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 28
Participants | 19 | 27

10. Secondary Outcome: Length of ICU Length of Stay
Description: Length of ICU stay in days, for participants who entered ICU
Time Frame: 28 days
Population: Analysis population is those participants in each group that entered the ICU
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 27 | 26
days | 17.59 (10.16) | 22.12 (10.37)

11. Secondary Outcome: Intensive Care Unit (ICU) Mortality
Description: Count of patients admitted to the ICU who die in ICU
Time Frame: 28 days
Population: Data was not collected or analyzed for this outcome
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Hospital Length of Stay
Description: Length of hospital stay in days
Time Frame: 28 days
Population: Data not available for 1 Group B participants
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 27
days | 23.63 (9.83) | 26.41 (11.12)

13. Secondary Outcome: Ventilator Free Days
Description: Number of ventilator-free hospitalized days
Time Frame: 28 days
Population: Data available in Group A for 8 of 15 participants who were intubated, and in Group B for 7 of 15 participants who were intubated
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 7
days | 9.13 (12.64) | 14.23 (14.80)

14. Secondary Outcome: Intubation Duration
Description: Length of intubation, measured in days
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 28
days | 4.12 (6.23) | 13.93 (9.45)

15. Secondary Outcome: Readmission
Description: Count of participants readmitted to hospital following index procedure hospital discharge
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 28
Participants | 6 | 3

16. Secondary Outcome: Serum Anti-SARS-CoV-2 IgG
Description: Count of participants positive for serum anti-SARS-CoV-2 IgG as assayed by the EUROIMMUN Anti-SARS-CoV-2 assay, evaluated semi-quantitatively by calculation of a ratio of the extinction of the patient sample over the extinction of a calibrator. This ratio is interpreted as: ratio < 0.8 is negative, ratio ≥ 0.8 to <1.0 is considered borderline, and ratio ≥ 1.1 is positive.
Time Frame: During hospitalization, a maximum of 28 days
Population: A change in the Emergency Use Authorization for plasma transfusion during COVID-19 occurred during the study. Untitered plasma was no longer available. Thus, data was not analyzed for this outcome.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: SARS-CoV-2 RNA
Description: Count of participants with presence of SARS-CoV-2 RNA detected by reverse transcription polymerase chain reaction (RT-PCR) tested nasopharyngeal swabs.
Time Frame: During hospitalization, a maximum of 28 days
Population: Data not available for 4 out of the 43 Group A participants. Data not available for 3 out of the 28 Group B participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 39 | 25
Participants | 36 | 22

18. Secondary Outcome: Mortality (Group A)
Description: Count of group A participants (non-intubated participants requiring >6 L supplemental oxygen to maintain oxygen saturation >92% at time of study entry and admitted <14 days) who die
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A
Number analyzed (Participants) | 43
Participants | 21

19. Secondary Outcome: Time From Transfusion to End of Ventilator Support (Group B)
Description: Number of days from transfusion date until end of ventilator support for surviving group B participants (participants who are intubated at study entry)
Time Frame: During hospitalization, a maximum of 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group B
Number analyzed (Participants) | 28
days | 6.25 (5.76)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 24/43 | 20/28
Serious Adverse Events (participants affected / at risk) | 24/43 | 20/28
Other Adverse Events (participants affected / at risk) | 3/43 | 4/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=43) | Group B (N=28)
Cardio-circulatory arrest (Cardiac disorders) | 1 (1) | 7 (7)
Neurological (Nervous system disorders) | 0 (0) | 3 (4)
Bleeding or low hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 21 (29) | 13 (16)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=43) | Group B (N=28)
pneumomediastinum (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Low hemaglobin (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Anterior rectal tear (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep right ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Minor allergic reaction (Immune system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to changes in the Emergency Use Authorization for plasma during COVID-19. All plasma was labeled either low titer or high titer. The protocol required untitered plasma be used, which resulted in inability to complete the study and early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT04432272/Prot_SAP_000.pdf